CLINICAL TRIAL: NCT02903186
Title: Multi-site Trial Using Short Mobile Messages (SMS) to Improve Infant Weight in Low-income Minorities
Brief Title: Multi-site Trial Using SMS to Improve Infant Weight
Acronym: SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Cristina Palacios, Associate Professor, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A4540315; 5U54MD008149-09 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-09-16 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: infants; minorities; overfeeding; WIC program; feeding practices; breastfeeding
MeSH Terms: conditions — Obesity; Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutrition messages (Experimental): The intervention will focus on reinforcing the WIC breastfeeding messages, preventing overfeeding (i.e. using spoon to feed baby, not adding baby food or cereal to bottle, not placing their babies to sleep with a bottle, feeding their babies without distractions, etc), delaying introduction of solid foods, and delaying and reducing baby juice consumption. Constructs in the transtheoretical model such as self-efficacy and decisional balance will be used to address key determinants of behavior change to ensure relevance to the audience, and will target individuals both at the earlier and later stages of change. The messages are written at a grade 5 level in Spanish (PR site) and English (Hawaii site) and will be sent on different days and times of the week.
  Interventions: Behavioral: SMS
- General health messages (Active Comparator): The control group will receive weekly SMS about general infant's health issues, such as placing the infant on his/her back to sleep, the timeline for immunizations, the proper use of car seats, asthma and other respiratory conditions common among small children, and other health information relevant to infants. The investigators will follow the same protocol (schedule, length, language, etc.) as for the intervention messages.
  Interventions: Behavioral: SMS

INTERVENTIONS:
Behavioral: SMS — This is an intervention using short mobile messages (SMS)

SUMMARY:
The goals of this multi-site clinical trial are to pilot test weekly SMS sent to parents/caregivers of infants to improve feeding practices and decrease excessive weight gain in infants who are participants of the Women, Infants and Children (WIC) program in Puerto Rico and Hawaii. The intervention consists of weekly SMS for 4 months to reinforce the feeding messages provided by WIC.

DETAILED DESCRIPTION:
The goals of this multi-site clinical trial are to pilot test weekly SMS sent to parents/caregivers of infants to improve feeding practices and decrease excessive weight gain in infants who are participants of the WIC program in two distinct locations, Puerto Rico and Hawaii; to assess acceptability and practicality of the intervention; and to assess acceptability of collecting blood spots in future studies. The investigators will recruit a convenience sample of parent/caregivers of infants 0-2 months participating in the WIC program in Puerto Rico and Hawaii to send weekly SMS for 4 months. The weekly messages will focus on reinforcing the breastfeeding messages provided by WIC, preventing overfeeding, delaying introduction of solid foods, and delaying and reducing baby juice consumption, which are key issues in low-income populations. Participants will complete validated questionnaires and anthropometry before and after the trial and results will be compared to the control group (no messages). Participants will also answer short questions by SMS at different points and an interview at the end of the trial to assess the SMS. The investigators will assess how many participants agree to collect blood spots in their infants in future studies.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver age 18 years and older
* owner of a mobile phone with unrestricted SMS capability
* responsible for the care of the infant and willing to actively participate for the full duration of the study.

Exclusion Criteria:

* infants with special diets
* infants with limited mobility
* pre-term birth (<37 weeks)
* small or large for gestational age (birthweight <10th or >90th p)
* inability to consent to participate in the study
* unwillingness to be randomized and not being able to read

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Excessive weight gain | 0-6 months
  Infant weight-for-length percentile will be calculated using the World Health Organization growth charts, as recommended by the Center for Disease Control and Prevention (CDC) for this age. Excessive weight will be categorized as ≥90th percentile

SECONDARY OUTCOMES:
Acceptability of collecting blood spots | 0-2 months
  When recruiting participants, the investigators will ask if they agree to participate in collecting a blood spot sample in their infants. This will be done through a short questionnaire.
Acceptability of the intervention - from short SMS | 0-6 months
  At different points of the trial, participants will be asked to answer short quantitative and qualitative questions sent by SMS about acceptability of the intervention. All answers to these questions will be summed and assign as "acceptable" if answers were positive 80% or greater of the times.
Acceptability of the intervention - from exit interview | 0-6 months
  Participants will complete a short semi-structured qualitative interview at the end of the trial to provide the opportunity to make open comments about the acceptability of the SMS. Answers from the interviews will be loaded into a qualitative data analysis software. Recordings will be transcribed verbatim for content analysis and the team will develop a coding scheme. Similar codes will be grouped into broader concepts to facilitate the analysis. Analysis will involve identifying recurring themes based.
Practicality of the intervention - from short SMS | 0-6 months
  At different points of the trial, participants will be asked to answer short quantitative and qualitative questions sent by SMS about practicality of the intervention. Answers will be summed and classified as "practical" if answers were positive 80% or greater of the times.
Practicality of the intervention - from exit interview | 0-6 months
  Participants will complete a short semi-structured qualitative interview at the end of the trial to provide the opportunity to make open comments about the practicality of the SMS. Answers from the interviews will be loaded into a qualitative data analysis software. Recordings will be transcribed verbatim for content analysis and the team will develop a coding scheme. Similar codes will be grouped into broader concepts to facilitate the analysis. Analysis will involve identifying recurring themes based.
Infant food frequency | 0-6 months
  This questionnaire includes 52 food items with a brief description on how these were prepared and/or their source (e.g., raw, canned, etc.). It also includes different portion sizes and information on supplements use. Using frequency of intake of each food and amount reported for each food, a total amount of each food per day will be calculated.
General infant feeding practices | 0-6 months
  This questionnaire includes questions about type of infant feeding (breast or bottle-feeding), type of milk used, age of stopping breastfeeding (exclusive and partial), age of introduction of juices and solid foods, use of the bottle to sleep baby, methods of feeding babies (i.e. using spoon, adding solids to bottle, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Palacios, PhD, Principal Investigator — Associate Professor
Locations (2):
- University of Hawaii at Manoa, Honolulu, Hawaii, United States
- University of Puerto Rico, Medical Sciences Campus (UPR-MSC), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Palacios C, Campos M, Gibby C, Melendez M, Lee JE, Banna J. Effect of a Multi-Site Trial using Short Message Service (SMS) on Infant Feeding Practices and Weight Gain in Low-Income Minorities. J Am Coll Nutr. 2018 Sep-Oct;37(7):605-613. doi: 10.1080/07315724.2018.1454353. Epub 2018 Apr 30. PMID 29708471
- [Result] Banna J, Campos M, Gibby C, Graulau RE, Melendez M, Reyes A, Lee JE, Palacios C. Multi-site trial using short mobile messages (SMS) to improve infant weight in low-income minorities: Development, implementation, lessons learned and future applications. Contemp Clin Trials. 2017 Nov;62:56-60. doi: 10.1016/j.cct.2017.08.011. Epub 2017 Aug 19. No abstract available. PMID 28827160
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Gibby CLK, Palacios C, Campos M, Graulau RE, Banna J. Acceptability of a text message-based intervention for obesity prevention in infants from Hawai'i and Puerto Rico WIC. BMC Pregnancy Childbirth. 2019 Aug 13;19(1):291. doi: 10.1186/s12884-019-2446-9. PMID 31409286
- [Derived] Gibby CLK, Palacios C, Campos M, Lim E, Banna J. Associations between gestational weight gain and rate of infancy weight gain in Hawai'i and Puerto Rico WIC participants. BMC Obes. 2018 Dec 3;5:41. doi: 10.1186/s40608-018-0219-z. eCollection 2018. PMID 30524746
- [Derived] Gibby CLK, Palacios C, Campos M, Lim E, Banna J. Breastfeeding Discontinuation Not Associated with Maternal Pregravid BMI But Associated with Native Hawaiian or Other Pacific Islander Race in Hawaii and Puerto Rico WIC Participants. Matern Child Health J. 2019 Jan;23(1):19-29. doi: 10.1007/s10995-018-2587-x. PMID 30006729